CLINICAL TRIAL: NCT01849809
Title: Safety and Effectiveness of Gamma Capsulotomy in Intractable Obsessive Compulsive Disorder
Brief Title: Safety and Effectiveness of Gamma Capsulotomy in Intractable OCD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Butler Hospital (Other)
Responsible Party: Principal Investigator, Steven Rasmussen, Medical Director, Butler Hospital, Butler Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB#2010-001
Record Dates: First submitted 2013-02-12; First posted 2013-05-09 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Obsessive Compulsive Disorder
MeSH Terms: conditions — Obsessive-Compulsive Disorder

STUDY DESIGN:
Masking Description: Open Label
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gamma Ventral Capsulotomy (Experimental)
  Interventions: Procedure: Gamma Ventral Capsulotomy

INTERVENTIONS:
Procedure: Gamma Ventral Capsulotomy

SUMMARY:
A research study of the effectiveness and safety of gamma knife ventral capsulotomy in patients with severe intractable obsessive-compulsive disorder (OCD).

ELIGIBILITY:
Inclusion Criteria:

1. OCD, diagnosed by Structured Clinical Interview for DSM-IV (SCID-IV), judged of disabling severity with a Yale-Brown Obsessive Compulsive Scale (YBOCS) score of at least 30 and a Social and Occupational Functioning Assessment Scale (SOFAS) score of 45 or less.
2. Persistence of severe symptoms and impairment for five or more years despite: 1. at least three adequate (≥3 months at the maximum tolerated dose) serotonin transporter inhibitor trials (fluoxetine, sertraline, fluvoxamine, paroxetine, citalopram, escitalopram, or clomipramine) alone or in combination with, 2. adequate behavior therapy (≥20 sessions of expert exposure and response prevention), and 3. augmentation of one of the selective SRIs with clomipramine, a neuroleptic, and clonazepam.
3. Age between 18 and 65 years.
4. Able to understand and comply with instructions.
5. Able to give fully informed, written consent in the judgment of the Consent Monitor.
6. Either drug free or on a stable drug regimen for at least 6 weeks.
7. Good general health.
8. A family member or significant other is available and willing to communicate with the research team if the patient's clinical status worsens.
9. The local referring psychiatrist is willing to provide ongoing care.

Exclusion Criteria:

1. Current or past psychotic disorder.
2. Full-scale IQ below 85.
3. A clinical history of bipolar mood disorder.
4. Any current clinically significant neurological disorder or medical illness affecting brain function, other than tic disorders or Tourette syndrome.
5. Any clinically significant abnormality on preoperative magnetic resonance imaging (MRI).
6. Inability to undergo presurgical MRI (cardiac pacemaker, pregnancy, metal in body, severe claustrophobia.
7. Current or unstably remitted substance abuse, dependence, or a positive urine toxicology screen.
8. Pregnancy and women of childbearing age not using effective contraception.
9. Unable to adhere to operational and administrative study requirements (in the investigators' judgment).
10. Clinical history of severe personality disorder.
11. Imminent risk of suicide (in the investigators' judgment).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 1993-02; Primary Completion 2011-08 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
Yale-Brown Obsessive Compulsive Severity Scale | Baseline to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Steven Rasmussen, MD, Principal Investigator — Butler Hospital
Locations (1):
- Butler Hospital, Providence, Rhode Island, United States

REFERENCES:
- [Derived] Rasmussen SA, Noren G, Greenberg BD, Marsland R, McLaughlin NC, Malloy PJ, Salloway SP, Strong DR, Eisen JL, Jenike MA, Rauch SL, Baer L, Lindquist C. Gamma Ventral Capsulotomy in Intractable Obsessive-Compulsive Disorder. Biol Psychiatry. 2018 Sep 1;84(5):355-364. doi: 10.1016/j.biopsych.2017.11.034. Epub 2017 Dec 15. PMID 29361268